CLINICAL TRIAL: NCT03199885
Title: A Randomized, Double-Blind, Phase III Trial of Taxane/Trastuzumab/Pertuzumab With Atezolizumab or Placebo in First-Line HER2-Positive Metastatic Breast Cancer
Brief Title: Testing the Drug Atezolizumab or Placebo With Usual Therapy in First-Line HER2-Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCI-2017-01119; NCI-2017-01119 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BR004 (Other: NRG Oncology); NRG-BR004 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2017-06-26; First posted 2017-06-27 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Breast Adenocarcinoma; Metastatic HER2-Positive Breast Carcinoma; Recurrent Breast Adenocarcinoma; Recurrent HER2-Positive Breast Carcinoma; Stage III Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7; Unresectable Breast Carcinoma; Unresectable HER2-Positive Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — atezolizumab; Biopsy; Docetaxel; Magnetic Resonance Spectroscopy; Paclitaxel; Taxes; pertuzumab; 2C4 antibody; Trastuzumab; CT-P6; PF-05280014; Ogivri; Ontruzant; trastuzumab biosimilar HLX02

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (pertuzumab, trastuzumab, taxane therapy, placebo) (Active Comparator): Patients receive pertuzumab IV over 30-60 minutes on days 1 and 22, trastuzumab IV over 30-90 minutes on days 1 and 22, and paclitaxel IV over 60 minutes on days 1, 8, 15, 22, 29, and 36 or docetaxel IV over 60 minutes on days 1 and 22. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive placebo IV 30-60 minutes on day 22 of cycle 1 and days 1 and 22 of subsequent cycles. Cycles repeat every 6 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a CT or MRI at baseline, prior to weeks 10, 19, 28 and then at 9, 12, 15, 18, 21, and 24 months from study entry, every 3 months through year 3, every 6 months for years 4 and 5, and then every 6 months for years 6 through 10 from study entry. Patients undergo a bone scan at baseline, every 6 months from study entry, every 6 months through year 3, and every 12 months for years 4 and 5.
  Interventions: Procedure: Biopsy; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Docetaxel; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Biological: Pertuzumab; Other: Placebo Administration; Other: Quality-of-Life Assessment; Biological: Trastuzumab
- Arm II (pertuzumab, trastuzumab, taxane therapy, atezolizumab) (Experimental): Patients receive pertuzumab, trastuzumab, and paclitaxel or docetaxel as in Arm I. Patients also receive atezolizumab IV over 30-60 minutes on day 22 of cycle 1 and days 1 and 22 of subsequent cycles. Cycles repeat every 6 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a CT or MRI at baseline, prior to weeks 10, 19, 28 and then at 9, 12, 15, 18, 21, and 24 months from study entry, every 3 months through year 3, every 6 months for years 4 and 5, and then every 6 months for years 6 through 10 from study entry. Patients undergo a bone scan at baseline, every 6 months from study entry, every 6 months through year 3, and every 12 months for years 4 and 5.
  Interventions: Drug: Atezolizumab; Procedure: Biopsy; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Docetaxel; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Biological: Pertuzumab; Other: Quality-of-Life Assessment; Biological: Trastuzumab

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
  Arms: Arm II (pertuzumab, trastuzumab, taxane therapy, atezolizumab)
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Pertuzumab — Given IV
  Other Names: 2C4; 2C4 Antibody; BCD-178; EG1206A; HLX11; HS627; MoAb 2C4; Monoclonal Antibody 2C4; Omnitarg; Perjeta; Pertuzumab Biosimilar BCD-178; Pertuzumab Biosimilar EG1206A; Pertuzumab Biosimilar HLX11; Pertuzumab Biosimilar HS627; Pertuzumab Biosimilar TQB2440; Rhumab 2C4; rhuMAb2C4; RO4368451; TQB 2440; TQB-2440; TQB2440
Other: Placebo Administration — Given IV
  Arms: Arm I (pertuzumab, trastuzumab, taxane therapy, placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; ALT02; Biceltis; CANMab; CT-P06; CT-P6; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Hercessi; Herclon; Hertraz; Herwenda; Herzuma; Kanjinti; Ogivri; Ontruzant; PF-05280014; QL 1701; QL-1701; QL1701; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; Trastuzumab Biosimilar CT-P6; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar QL1701; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-herw; Trastuzumab-pkrb; Trastuzumab-qyyp; Trastuzumab-strf; Trastuzumab-zerc; Trazimera; Zercepac

SUMMARY:
This randomized phase III trial studies how well paclitaxel, trastuzumab, and pertuzumab with or without atezolizumab works in treating patients with breast cancer that has spread to other parts of the body (metastatic). Chemotherapy drugs, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Trastuzumab is a form of "targeted therapy" because it works by attaching itself to specific molecules (receptors) on the surface of cancer cells, known as HER2 receptors. When trastuzumab attaches to HER2 receptors, the signals that tell the cells to grow are blocked and the cancer cell may be marked for destruction by the body's immune system. Monoclonal antibodies, such as pertuzumab, may interfere with the ability of cancer cells to grow and spread. Immunotherapy with monoclonal antibodies, such as atezolizumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. It is not yet known whether giving paclitaxel, trastuzumab, and pertuzumab with or without atezolizumab may kill more tumor cells.

*NOTE: This study has a central confirmation step. The purpose of this step is to confirm by central testing that the patient's tumor has specific receptors. If the patient meets all the study requirements, the patient will join the study and begin therapy for breast cancer while the tumor is being tested.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether the addition of atezolizumab to a regimen of pertuzumab and trastuzumab combined with a taxane (paclitaxel or docetaxel) will improve the progression-free survival (PFS), assessed by investigator using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, relative to the addition of a placebo to a regimen of pertuzumab and trastuzumab combined with a taxane (paclitaxel or docetaxel) in patients with newly documented HER2-positive measurable metastatic breast cancer.

SECONDARY OBJECTIVES:

I. To determine whether the addition of atezolizumab to a regimen of pertuzumab and trastuzumab combined with a taxane (paclitaxel or docetaxel) will improve the overall survival (OS) relative to the addition of placebo to a regimen of pertuzumab and trastuzumab, combined with a taxane (paclitaxel or docetaxel).

II. To determine whether the addition of atezolizumab to a regimen of pertuzumab and trastuzumab combined with a taxane (paclitaxel or docetaxel) will improve the overall objective response (OR) in the cohort of patients randomized 6 months or more prior to study accrual closure assessed by investigator using RECIST 1.1 criteria, relative to the addition of placebo to a regimen of pertuzumab and trastuzumab combined with a taxane (paclitaxel or docetaxel).

III. To determine the immune-related toxicity profile of the two treatment regimens.

IV. To determine the cardiac safety profile of the two treatment regimens.

EXPLORATORY OBJECTIVES:

I. To determine whether the addition of atezolizumab to a regimen of pertuzumab and trastuzumab combined with a taxane (paclitaxel or docetaxel) will decrease the incidence of subsequent brain metastases in patients without known brain metastases at study entry relative to the addition of a placebo to a regimen of pertuzumab and trastuzumab combined with a taxane (paclitaxel or docetaxel).

II. To determine the utility of PD-L1 immunohistochemistry (IHC) staining as a predictive and prognostic biomarker associated with clinical response, as assessed by investigator using RECIST 1.1 criteria, to atezolizumab in combination with trastuzumab and pertuzumab combined with a taxane (paclitaxel or docetaxel).

III. To identify potential biomarkers that can predict benefit from the addition of atezolizumab in patients with newly documented HER2-positive measurable metastatic breast cancer treated with a regimen of pertuzumab and trastuzumab combined with a taxane (paclitaxel or docetaxel).

IV. To explore the toxicity profile of the two treatment regimens using patient-reported symptomatic adverse events in addition to standard adverse event reports.

V. To determine the feasibility and added value of frequent assessment of toxicity using Patient Reported Outcomes (PRO)-Common Terminology Criteria for Adverse Events (CTCAE) with electronic(e)PRO reporting.

VI. To explore whether the addition of atezolizumab to a regimen of pertuzumab and trastuzumab combined with a taxane (paclitaxel or docetaxel) will contribute to increased patient-reported fatigue in comparison to the addition of placebo to a regimen of pertuzumab and trastuzumab combined with a taxane (paclitaxel or docetaxel).

OUTLINE:

STEP 1: Patients receive pertuzumab intravenously (IV) over 30-60 minutes on days 1 and 22, trastuzumab IV over 30-90 minutes on days 1 and 22, and paclitaxel IV over 60 minutes on days 1, 8, 15, 22, 29, and 36 or docetaxel IV over 60 minutes on days 1 and 22. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients may undergo a biopsy at baseline. Patients undergo computed tomography (CT), magnetic resonance imaging (MRI), and/or bone scan at baseline.

STEP 2: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive pertuzumab IV over 30-60 minutes on days 1 and 22 of each cycle, trastuzumab IV over 30-90 minutes on days 1 and 22 of each cycle, and paclitaxel IV over 60 minutes on days 1, 8, 15, 22, 29, and 36 of each cycle or docetaxel IV over 60 minutes on days 1 and 22 of each cycle. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive atezolizumab IV over 30-60 minutes on day 22 of cycle 1 and days 1 and 22 of subsequent cycles. Cycles repeat every 6 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a CT or MRI at baseline, prior to weeks 10, 19, 28 and then at 9, 12, 15, 18, 21, and 24 months from study entry, every 3 months through year 3, every 6 months for years 4 and 5, and then every 6 months for years 6 through 10 from study entry. Patients undergo a bone scan at baseline, every 6 months from study entry, every 6 months through year 3, and every 12 months for years 4 and 5.

ARM II: Patients receive pertuzumab, trastuzumab, and paclitaxel or docetaxel as in Arm I. Patients also receive placebo IV 30-60 minutes on day 22 of cycle 1 and days 1 and 22 of subsequent cycles. Cycles repeat every 6 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a CT or MRI at baseline, prior to weeks 10, 19, 28 and then at 9, 12, 15, 18, 21, and 24 months from study entry, every 3 months through year 3, every 6 months for years 4 and 5, and then every 6 months for years 6 through 10 from study entry. Patients undergo a bone scan at baseline, every 6 months from study entry, every 6 months through year 3, and every 12 months for years 4 and 5.

After completion of study treatment, patients are followed up at 30 days and every 3 months for 3 years and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have signed and dated an Institutional Review Board (IRB)-approved consent form that conforms to federal and institutional guidelines
* The trial is open to female and male patients
* Patients must be >= 18 years old
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically confirmed adenocarcinoma of the breast with locally recurrent, unresectable disease or metastatic disease outside the central nervous system (CNS) confirmed as described below; eligible patients include those with either:

  * De novo metastatic disease presenting without prior history of HER2-positive breast cancer:

    * Diagnosis should have been made from a biopsy of a metastatic disease site, but biopsy from the breast primary or involved regional lymph nodes is acceptable if biopsy of the metastatic sites was thought to carry excessive risk for the patient
  * Locally recurrent or metastatic disease following prior therapy for early breast cancer:

    * Diagnosis must have been made from the biopsy of the locally recurrent or metastatic disease
    * There must be an interval of >= 6 months between completion of neoadjuvant/adjuvant HER2-targeted therapy and documentation of locally recurrent or metastatic HER2-positive disease by biopsy
* Patients must have measurable disease based on RECIST 1.1, as determined by the site, which has not been irradiated to be eligible
* Patients with brain metastases are eligible if they meet ALL the following criteria:

  * Four or fewer metastatic sites to CNS
  * Largest unexcised tumor does not exceed 3 cm
  * No metastases to brain stem, midbrain, pons, medulla or the optic nerves and chiasm
  * Must have measurable disease outside the CNS, based on RECIST 1.1, as determined by the site, which has not been irradiated
  * If patient presented with symptoms from CNS metastases, the symptoms must have resolved with initiation of steroids and initial local therapy (surgery, radiation therapy, or both)
  * Must have been evaluated by Medical Oncologist and plan is to administer trastuzumab, pertuzumab, and a taxane as first-line systemic therapy
  * May have received administration of trastuzumab OR lapatinib concurrently with radiation therapy for brain metastases. Toxicities related to lapatinib if administered, should be =< grade 1 per the CTCAE v5.0, and the lapatinib must have been completed at least 2 weeks prior to study entry
  * No history of intracranial hemorrhage or spinal cord hemorrhage
  * No neurosurgical resection or brain biopsy within 10 days prior to study entry
* After study entry and before randomization, send tissue for central HER2 confirmation; a tumor specimen obtained at the time of diagnosis of locally recurrent or metastatic disease must have been determined to be HER2-positive based on local testing according to American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines (Wolff 2018); HER2 status should initially be assessed using an Food and Drug Administration (FDA)-cleared IHC assay; positive is defined as IHC 3+ staining intensity; if HER2 IHC results are equivocal (2+), then HER2 status will be determined using a FDA-cleared HER2 in situ hybridization (ISH) test according to ASCO/CAP guidelines; Note: Once HER2-positive is confirmed on central testing, patients will be randomized to atezolizumab/placebo; randomization within 14 days from study entry will ensure that the Pharmaceutical Management Branch (PMB)-supplied agents will be received at the site for treatment on day 22 of cycle 1
* The tumor specimen obtained at the time of diagnosis used for HER2 testing must also have central testing for PD-L1 status; patients will be eligible irrespective of PD-L1 testing result including PD-L1 indeterminant
* The tumor specimen obtained at the time of diagnosis used for HER2 and PD-L1 testing should also have central testing for estrogen receptor (ER) and progesterone receptor (PgR) according to current ASCO/CAP guideline recommendations for hormone receptor testing; patients with < 1% ER and PgR staining by IHC will be classified as negative; if enough material for central confirmation of ER and PgR is unavailable, local testing results for ER and PgR may be used for eligibility
* Localized palliative radiation therapy to sites of non-measurable disease is allowed for symptom management and may begin prior to study entry and continue following study entry while receiving study therapy
* Patients must have imaging of the chest/abdomen/pelvis, preferably with a CT scan, and a bone scan within 5 weeks prior to study entry; (NOTE: if a patient is unable to receive CT contrast, a MRI of the abdomen/pelvis and non-contrast chest CT should be performed; positron emission tomography/computed tomography [PET/CT] is not an acceptable alternative)
* MRI of the brain (or contrast CT scan of the brain if patients are unable to undergo MRI) must be obtained in patients with symptoms suggesting possible central nervous system (CNS) metastatic disease; neuroimaging is recommended but not required in asymptomatic patients
* Absolute neutrophil count (ANC) must be >= 1200/mm^3 (within 14 days prior to study entry)
* Platelet count must be >= 100,000/mm^3 (within 14 days prior to study entry)
* Hemoglobin must be >= 8 g/dL (within 14 days prior to study entry)
* Total bilirubin must be =< 1.5 x upper limit of normal (ULN) for the lab or direct bilirubin =< ULN for patients with bilirubin levels > 1.5 x ULN (within 14 days prior to study entry)
* Aspartate aminotransferase (AST) and alanine aminotransaminase (ALT) must be =< 2.5 x ULN for the lab or =< 5 x ULN for patients with liver metastases (within 14 days prior to study entry)
* Serum creatinine =< 1.5 x ULN or measured or calculated creatinine clearance >= 50 mL/min using the Cockcroft-Gault formula for patients with creatinine levels > 1.5 x ULN for the lab (within 14 days prior to study entry)
* Patients not receiving anti-coagulant therapy must have prothrombin time (PT) and international normalized ratio (INR) =< 1.5 x ULN within 14 days prior to study entry; for laboratories that do not report an ULN for the INR assay, use =< 1.5 as the value for the ULN; patients receiving anti-coagulants should have a baseline INR assessed, but the value does not affect eligibility
* A serum thyroid-stimulating hormone (TSH) and AM (preferably in morning) cortisol must be obtained within 14 days prior to study entry to obtain a baseline value; patients with abnormal TSH or AM cortisol baseline levels should be further evaluated and managed per institutional standards; asymptomatic patients who require initiation or adjustment of medication or are followed without initiating treatment based on endocrinologist's recommendations are eligible
* Left ventricular ejection fraction (LVEF) assessment must be performed within 6 weeks prior to study entry; (LVEF assessment performed by echocardiogram is preferred; however, multigated acquisition scan (MUGA) scan may be substituted based on institutional preferences); the LVEF must be >= 50% regardless of the cardiac imaging facility's lower limit of normal
* Administration of atezolizumab may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality; women of child-bearing potential and men must agree to use adequate contraception (non-hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 5 months (150 days) after the last dose of atezolizumab/placebo and 7 months after the last dose of trastuzumab and pertuzumab; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of study entry are eligible for this trial

Exclusion Criteria:

* Patients with brain metastases are excluded if they meet ANY of the following criteria:

  * Symptoms from brain metastases have not resolved prior to study entry
  * Five or more clearly identified foci of metastases to the brain
  * Largest unexcised tumor exceeds 3 cm
  * Spinal cord metastases
  * Medical Oncologist plans to employ HER2-directed tyrosine kinase inhibitor as component of systemic therapy
  * Metastatic disease limited to CNS
* Leptomeningeal carcinomatosis
* History of systemic anti-cancer therapy (e.g., chemotherapy, targeted therapy) for metastatic breast cancer (MBC) except as described in inclusion criteria
* History of exposure to cumulative doses of doxorubicin greater than 360 mg per square meter of body-surface area or its equivalent
* Prior treatment with mTOR inhibitors or CDK 4/6 inhibitors in combination with endocrine therapy for treatment of metastatic disease
* Prior treatment with CD137 agonists or immune checkpoint-blockade therapies, including anti-CD40, anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* History of non-breast malignancies (except for in situ cancers treated only by local excision and basal cell and squamous cell carcinomas of the skin) within 5 years prior to study entry
* Uncontrolled hypertension defined as sustained systolic blood pressure (BP) > 150 mmHg or diastolic BP > 90 mmHg; (patients with initial BP elevations are eligible if initiation or adjustment of BP medication lowers pressure to meet entry criteria)
* History of asymptomatic LVEF decline to < 40% during or after prior HER2-targeted therapy even if the current LVEF is >= 50%
* Cardiac disease (history of and/or active disease) that would preclude the use of the drugs included in the treatment regimens; this includes but is not confined to:

  * Active cardiac disease

    * Angina pectoris that requires the current use of anti-anginal medication;
    * Ventricular arrhythmias except for benign premature ventricular contractions;
    * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication;
    * Conduction abnormality requiring a pacemaker;
    * Valvular disease with documented compromise in cardiac function; or
    * Symptomatic pericarditis
  * History of cardiac disease

    * Prior myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular (LV) function;
    * History of documented congestive heart failure (CHF) defined as symptomatic heart failure with an LVEF < 40%; or
    * Documented cardiomyopathy
* Nervous system disorder (paresthesia, peripheral motor neuropathy, or peripheral sensory neuropathy) >= grade 2, per the CTCAE v 5.0
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to pertuzumab or trastuzumab or to any of its excipients, as well as any chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or other recombinant antibodies
* Known allergy or hypersensitivity to the components of the atezolizumab formulation or to any of the study drugs or excipients, (e.g., Cremophor EL, polysorbate 80)
* History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low-potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying conditions within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* Treatment with systemic immunomodulatory medications (including but not limited to interferons, IL-2) within 4 weeks or 5 half-lives of the drug, whichever is longer, prior to study entry
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis [anti-TNF] factor agents) within 14 days prior to study entry or anticipation of need for systemic immunosuppressive medications during the study; Note: Intranasal and inhaled corticosteroids or systemic corticosteroids at doses that do not exceed 10 mg/day of prednisone or an equivalent corticosteroid are allowed
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 2 weeks prior to study entry
* Active hepatitis B virus (HBV) infection, defined as having a positive hepatitis B surface antigen (HBsAg) test at screening; patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test at screening, are eligible for the study if active HBV infection is ruled out on the basis of HBV deoxyribonucleic acid (DNA) viral load per local guidelines
* Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test at screening confirmed by a polymerase chain reaction (PCR) positive for HCV ribonucleic acid (RNA)
* Patients with clinically active tuberculosis
* Severe infection within 4 weeks prior to study entry, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Prior allogeneic stem cell or solid organ transplantation
* Symptomatic peripheral ischemia
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis or >= grade 1 pulmonary fibrosis, per the CTCAE v5.0, on screening chest CT scan
* Administration of a live, attenuated vaccine within 4 weeks prior to study entry or anticipation that such vaccine will be required during the study

  * Patients must agree not to receive live, attenuated influenza vaccine (e.g., FluMist) within 4 weeks prior to study entry, during treatment or within 5 months following the last dose of atezolizumab/placebo
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements or interfere with interpretation of study results
* Pregnancy or lactation at the time of study entry or intention to become pregnant during the study; (Note: Pregnancy testing according to institutional standards for women of childbearing potential must be performed within 3 days prior to study entry)
* Use of any investigational product within 4 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles E Geyer, Principal Investigator — NRG Oncology
Locations (673):
- United States (662):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Katmai Oncology Group, Anchorage, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - Banner Boswell Medical Center, Sun City, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - City of Hope South Bay, Torrance, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - GenesisCare USA - Aventura FP, Aventura, Florida
  - GenesisCare USA - Boca Ration FP06, Boca Raton, Florida
  - AdventHealth Celebration, Celebration, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta Oncology Associates PC-D'Antignac, Augusta, Georgia
  - Augusta Oncology Associates PC-Wheeler, Augusta, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Eisenhower Army Medical Center, Fort Eisenhower, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Piedmont Newnan Hospital, Newnan, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Suburban Hematology Oncology Associates - Snellville, Snellville, Georgia
  - Piedmont Henry Hospital, Stockbridge, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Mission Cancer and Blood - West Des Moines, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Medical Oncology, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Waldo County General Hospital, Belfast, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - FMH James M Stockman Cancer Institute, Frederick, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Kensington Medical Center, Kensington, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Cancer Partners of Nebraska - Pine Lake, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Neurosurgeons of New Jersey-Ridgewood, Ridgewood, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Valley Medical Group - Wayne Multispecialty Practice, Wayne, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Good Samaritan University Hospital, West Islip, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Messino Cancer Centers, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Atrium Health Lincoln/LCI-Lincolnton, Lincolnton, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Nash UNC HealthCare, Rocky Mount, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - Crozer Regional Cancer Center at Brinton Lake, Glen Mills, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Redeemer Health, Meadowbrook, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Crozer-Chester Medical Center, Upland, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Thompson Cancer Survival Center - West, Knoxville, Tennessee
  - Thompson Oncology Group-Lenoir City, Lenoir City, Tennessee
  - Thompson Oncology Group-Maryville, Maryville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Thompson Oncology Group-Oak Ridge, Oak Ridge, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Wellmont Medical Associates-Bristol, Bristol, Virginia
  - Kaiser Permanente-Burke Medical Center, Burke, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (11):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA-Vancouver Island Cancer Centre, Victoria, British Columbia
  - The Moncton Hospital, Moncton, New Brunswick
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - William Osler Health System-Brampton Civic Hospital, Brampton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Algoma District Cancer Program Sault Area Hospital, Sault Ste. Marie, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CSSS Champlain-Charles Le Moyne, Greenfield Park, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Bandos H, Kim S, Henry NL, Hays RD, Calsavara VF, Luu M, Gresham G, Lu KY, Irvin WJ Jr, Suga JM, Siddique S, Cecchini RS, Rogatko A, Yothers G, Tighiouart M, Ganz PA. Feasibility of frequent monitoring of symptoms using the PRO-CTCAE in the NRG-BR004 clinical trial. JNCI Cancer Spectr. 2025 Apr 30;9(3):pkaf032. doi: 10.1093/jncics/pkaf032. PMID 40170372

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Pertuzumab, Trastuzumab, Taxane Therapy, Placebo): Patients receive pertuzumab IV over 30-60 minutes on days 1 and 22, trastuzumab IV over 30-90 minutes on days 1 and 22, and paclitaxel IV over 60 minutes on days 1, 8, 15, 22, 29, and 36 or docetaxel IV over 60 minutes on days 1 and 22. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive placebo IV 30-60 minutes on day 22 of cycle 1 and days 1 and 22 of subsequent cycles. Cycles repeat every 6 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a CT or MRI at baseline, prior to weeks 10, 19, 28 and then at 9, 12, 15, 18, 21, and 24 months from study entry, every 3 months through year 3, every 6 months for years 4 and 5, and then every 6 months for years 6 through 10 from study entry. Patients undergo a bone scan at baseline, every 6 months from study entry, every 6 months through year 3, and every 12 months for years 4 and 5.
  Biopsy: Undergo biopsy Bone Scan: Undergo bone scan Computed Tomography: Undergo CT scan Docetaxel: Given IV Magnetic Resonance Imaging: Undergo MRI Paclitaxel: Given IV Pertuzumab: Given IV Placebo Administration: Given IV Quality-of-Life Assessment: Ancillary studies Trastuzumab: Given IV
- Arm II (Pertuzumab, Trastuzumab, Taxane Therapy, Atezolizumab): Patients receive pertuzumab, trastuzumab, and paclitaxel or docetaxel as in Arm I. Patients also receive atezolizumab IV over 30-60 minutes on day 22 of cycle 1 and days 1 and 22 of subsequent cycles. Cycles repeat every 6 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a CT or MRI at baseline, prior to weeks 10, 19, 28 and then at 9, 12, 15, 18, 21, and 24 months from study entry, every 3 months through year 3, every 6 months for years 4 and 5, and then every 6 months for years 6 through 10 from study entry. Patients undergo a bone scan at baseline, every 6 months from study entry, every 6 months through year 3, and every 12 months for years 4 and 5.
  Atezolizumab: Given IV Biopsy: Undergo biopsy Bone Scan: Undergo bone scan Computed Tomography: Undergo CT scan Docetaxel: Given IV Magnetic Resonance Imaging: Undergo MRI Paclitaxel: Given IV Pertuzumab: Given IV Quality-of-Life Assessment: Ancillary studies Trastuzumab: Given IV
Period: Overall Study
Arm/Group | Arm I (Pertuzumab, Trastuzumab, Taxane Therapy, Placebo) | Arm II (Pertuzumab, Trastuzumab, Taxane Therapy, Atezolizumab)
Started | 93 | 97
Completed | 70 | 72
Not Completed | 23 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Pertuzumab, Trastuzumab, Taxane Therapy, Placebo) | Arm II (Pertuzumab, Trastuzumab, Taxane Therapy, Atezolizumab) | Total
Number analyzed (Participants) | 93 | 97 | 190
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 77 | 151
  >=65 years | 19 | 20 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 96 | 186
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 8 | 21
  Not Hispanic or Latino | 77 | 85 | 162
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 3 | 8 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 8 | 11 | 19
  White | 76 | 70 | 146
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Will be determined using the current Response Evaluation Criteria in Solid Tumors 1.1 criteria. Analysis will be based on the intent to treat population. The stratified log-rank test will be used to compare the progression free survival between the two treatment arms with the following stratification factors: prior neoadjuvant or adjuvant therapy with trastuzumab (no; yes), estrogen receptor status (positive; negative), disease sites (any visceral without brain metastasis; non-visceral only without brain metastasis; brain metastasis), and choice of taxane (paclitaxel; docetaxel). The Kaplan-Meier estimates will be calculated by treatment arms. Stratified Cox proportional hazards models to estimate the hazard ratio.
Time Frame: At the definitive analysis 2.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Pertuzumab, Trastuzumab, Taxane Therapy, Placebo) | Arm II (Pertuzumab, Trastuzumab, Taxane Therapy, Atezolizumab)
Number analyzed (Participants) | 93 | 97
percentage of participants | 40.5 [29.7 to 51.0] | 52.3 [41.4 to 62.2]

2. Secondary Outcome: Overall Survival (OS)
Description: Analysis will be based on the intent to treat population. The stratification factors are the same as what are used in the stratified log-rank test for the primary analysis on progression free survival. The Kaplan-Meier estimates will be calculated by treatment arms. Stratified Cox proportional hazards models to estimate the hazard ratio.
Time Frame: At definitive analysis-2.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Pertuzumab, Trastuzumab, Taxane Therapy, Placebo) | Arm II (Pertuzumab, Trastuzumab, Taxane Therapy, Atezolizumab)
Number analyzed (Participants) | 93 | 97
percentage of participants | 86.3 [77.5 to 93.0] | 87.4 [77.1 to 92.1]

3. Secondary Outcome: Overall Objective Response
Description: Defined as complete response or partial response. Will be determined using Response Evaluation Criteria in Solid Tumors 1.1 criteria. The stratified Cochran-Mantel-Haenszel test will be used to compare the object response between the treatment arms.
Time Frame: 38 months after study activation.
Population: This analysis was restricted to the sub-cohort of patients randomized six months or more prior to May 20, 2022. Only response data collected up to May 20, 2022, were included in this analysis. We used RECIST v1.1. It involves target lesion, nontarget lesion, second primary cancer, and death.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Pertuzumab, Trastuzumab, Taxane Therapy, Placebo) | Arm II (Pertuzumab, Trastuzumab, Taxane Therapy, Atezolizumab)
Number analyzed (Participants) | 77 | 68
percentage of participants | 79.4 [68.4 to 87.3] | 77.9 [67.5 to 85.7]

4. Secondary Outcome: Frequency of Adverse Events, Including Late Immune-related Toxicities
Description: Will be categorized using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0. Comparisons of the adverse events between the two treatment arms will be done by the Fisher's exact test.
Time Frame: Every 6 months up to 8 years
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: 38 months from study activation.
Description: Participants at Risk includes any patient who submitted an AE form. Adverse event data were reported by sites on 187 patients. Some patients withdrew consent shortly after randomization and adverse event data were not submitted. However, they were still at risk for mortality prior to consent withdrawal. Therefore we did not have any data on adverse events from 3 BR004 participants. This led to the difference between the number at risk for mortality and number at risk for adverse events.
Groups:
- Arm I (Pertuzumab, Trastuzumab, Taxane Therapy, Placebo): Arm I (pertuzumab, trastuzumab, taxane therapy, placebo)
- Arm II (Pertuzumab, Trastuzumab, Taxane Therapy, Atezolizumab): Arm II (pertuzumab, trastuzumab, taxane therapy, atezolizumab)
Arm/Group | Arm I (Pertuzumab, Trastuzumab, Taxane Therapy, Placebo) | Arm II (Pertuzumab, Trastuzumab, Taxane Therapy, Atezolizumab)
All-Cause Mortality (participants affected / at risk) | 17/93 | 14/97
Serious Adverse Events (participants affected / at risk) | 24/91 | 27/96
Other Adverse Events (participants affected / at risk) | 90/91 | 96/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Pertuzumab, Trastuzumab, Taxane Therapy, Placebo) (N=91) | Arm II (Pertuzumab, Trastuzumab, Taxane Therapy, Atezolizumab) (N=96)
Adrenal insufficiency (Endocrine disorders) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 3
Alkaline phosphatase increased (Investigations) | 0 | 1
Anaphylaxis (Immune system disorders) | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac troponin T increased (Investigations) | 1 | 0
Catheter related infection (Infections and infestations) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 1 | 3
Creatinine increased (Investigations) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4
Fever (General disorders) | 2 | 2
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Heart failure (Cardiac disorders) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 3
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Immune system disorders - Other, specify (Immune system disorders) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 | 1
Kidney infection (Infections and infestations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 4
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Presyncope (Nervous system disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 1
Renal calculi (Renal and urinary disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Sepsis (Infections and infestations) | 2 | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0
Skin infection (Infections and infestations) | 2 | 2
Sudden death NOS (General disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 2 | 3
Urinary tract infection (Infections and infestations) | 0 | 2
Vasculitis (Vascular disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
White blood cell decreased (Investigations) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Enterocolitis infectious (Infections and infestations) | 2 | 1
Lung infection (Infections and infestations) | 2 | 4
Mitral valve disease (Cardiac disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Gallbladder infection (Infections and infestations) | 0 | 1
Hypophysitis (Endocrine disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 4
Pregnancy loss (Pregnancy, puerperium and perinatal conditions) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Pertuzumab, Trastuzumab, Taxane Therapy, Placebo) (N=91) | Arm II (Pertuzumab, Trastuzumab, Taxane Therapy, Atezolizumab) (N=96)
Abdominal pain (Gastrointestinal disorders) | 18 | 15
Adrenal insufficiency (Endocrine disorders) | 9 | 10
Alanine aminotransferase increased (Investigations) | 19 | 28
Alkaline phosphatase increased (Investigations) | 22 | 20
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 47 | 52
Anemia (Blood and lymphatic system disorders) | 55 | 59
Anorexia (Metabolism and nutrition disorders) | 26 | 31
Anxiety (Psychiatric disorders) | 11 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 13
Aspartate aminotransferase increased (Investigations) | 19 | 28
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 14
Bloating (Gastrointestinal disorders) | 6 | 2
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 5 | 10
Blood bilirubin increased (Investigations) | 2 | 9
Blurred vision (Eye disorders) | 8 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Breast pain (Reproductive system and breast disorders) | 6 | 6
Chills (General disorders) | 6 | 12
Colitis (Gastrointestinal disorders) | 4 | 7
Constipation (Gastrointestinal disorders) | 30 | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 26
Creatinine increased (Investigations) | 10 | 17
Dehydration (Metabolism and nutrition disorders) | 5 | 14
Depression (Psychiatric disorders) | 11 | 7
Diarrhea (Gastrointestinal disorders) | 72 | 82
Dizziness (Nervous system disorders) | 17 | 12
Dry eye (Eye disorders) | 9 | 4
Dry mouth (Gastrointestinal disorders) | 6 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 16 | 16
Dysgeusia (Nervous system disorders) | 19 | 23
Dyspepsia (Gastrointestinal disorders) | 11 | 13
Dysphagia (Gastrointestinal disorders) | 1 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 | 20
Dysuria (Renal and urinary disorders) | 7 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 26 | 24
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 | 9
Eye disorders - Other, specify (Eye disorders) | 10 | 12
Fatigue (General disorders) | 60 | 68
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 7
Fever (General disorders) | 12 | 11
Flu like symptoms (General disorders) | 12 | 10
Flushing (Vascular disorders) | 9 | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 7 | 7
General disorders and administration site conditions - Other, specify (General disorders) | 8 | 9
Generalized edema (General disorders) | 5 | 4
Headache (Nervous system disorders) | 28 | 28
Hemorrhoids (Gastrointestinal disorders) | 4 | 7
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 7 | 4
Hot flashes (Vascular disorders) | 24 | 16
Hyperglycemia (Metabolism and nutrition disorders) | 36 | 37
Hypertension (Vascular disorders) | 20 | 23
Hyperthyroidism (Endocrine disorders) | 5 | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 21 | 27
Hypocalcemia (Metabolism and nutrition disorders) | 12 | 27
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 6
Hypokalemia (Metabolism and nutrition disorders) | 27 | 33
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 12
Hyponatremia (Metabolism and nutrition disorders) | 20 | 25
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 5
Hypotension (Vascular disorders) | 6 | 5
Hypothyroidism (Endocrine disorders) | 6 | 18
Infections and infestations - Other, specify (Infections and infestations) | 30 | 24
Insomnia (Psychiatric disorders) | 28 | 23
Investigations - Other, specify (Investigations) | 8 | 5
Lymphocyte count decreased (Investigations) | 28 | 22
Memory impairment (Nervous system disorders) | 3 | 5
Mucositis oral (Gastrointestinal disorders) | 25 | 25
Muscle cramp (Musculoskeletal and connective tissue disorders) | 7 | 10
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 5 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 9
Nail changes (Skin and subcutaneous tissue disorders) | 16 | 18
Nail discoloration (Skin and subcutaneous tissue disorders) | 9 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Nausea (Gastrointestinal disorders) | 43 | 54
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 8
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 5
Neutrophil count decreased (Investigations) | 30 | 35
Pain (General disorders) | 17 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 12
Paresthesia (Nervous system disorders) | 12 | 14
Paronychia (Infections and infestations) | 5 | 2
Peripheral motor neuropathy (Nervous system disorders) | 6 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 53 | 56
Platelet count decreased (Investigations) | 4 | 8
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 23
Rash acneiform (Skin and subcutaneous tissue disorders) | 24 | 26
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 31 | 38
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Sinus tachycardia (Cardiac disorders) | 11 | 7
Sinusitis (Infections and infestations) | 6 | 6
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 19 | 19
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 5
Skin infection (Infections and infestations) | 9 | 10
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 | 13
Thromboembolic event (Vascular disorders) | 4 | 6
Upper respiratory infection (Infections and infestations) | 7 | 6
Urinary tract infection (Infections and infestations) | 12 | 14
Vomiting (Gastrointestinal disorders) | 22 | 33
Watering eyes (Eye disorders) | 5 | 6
Weight gain (Investigations) | 6 | 4
Weight loss (Investigations) | 16 | 17
White blood cell decreased (Investigations) | 31 | 39
Nail loss (Skin and subcutaneous tissue disorders) | 4 | 5
Edema limbs (General disorders) | 23 | 26
Ejection fraction decreased (Investigations) | 6 | 6
Infusion related reaction (Injury, poisoning and procedural complications) | 17 | 27
Lung infection (Infections and infestations) | 4 | 5
Nail infection (Infections and infestations) | 6 | 5
Non-cardiac chest pain (General disorders) | 2 | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 | 8
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT03199885/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT03199885/ICF_001.pdf